CLINICAL TRIAL: NCT05340751
Title: The Effect of Hypotensive Anesthesia on Hemoglobin Levels During Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-081
Record Dates: First submitted 2018-11-23; First posted 2022-04-22 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia
Keywords: Blood management; Blood transfusion; Hemoglobin; Hypotensive Anesthesia; Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anesthesia: hemoglobin
  Interventions: Diagnostic Test: Blood drawn

INTERVENTIONS:
Diagnostic Test: Blood drawn — Hemoglobin and Hematocrit Levels

SUMMARY:
The current study investigates the effect of hypotensive anesthesia on patient hemoglobin levels during primary total knee arthroplasty. Considering that because of the tourniquet there is no blood loss during the first 60 minutes of the procedure changes in hemoglobin during the first 60 minutes should be primarily related to decrease in blood pressure and secondary to fluid loading during hypotensive anesthesia.

DETAILED DESCRIPTION:
The specific aim of this prospective study is to collect serial hemoglobin levels intraoperatively during hypotensive anesthesia to evaluate if intraoperative intravenous fluid substitution will change hemoglobin levels during the time the tourniquet is inflated (no blood loss).

The combination of vasodilation during hypotensive anesthesia and fluid substitution will result in decrease of hemoglobin levels during the tourniquet time.

Tubes of 5cc to measure hemoglobin and hematocrit levels preoperatively, prior to inflation of the tourniquet, 15 minutes, 30 minutes, 45 minutes and 60 minutes after tourniquet inflation and in PACU as well as POD 1.

ELIGIBILITY:
Inclusion Criteria:

* Non- inflammatory degenerative joint disease of the knee
* Patients scheduled for unilateral primary total Knee arthroplasty
* Age between 40 and 80 years
* Hypotensive spinal-epidural anesthesia with systolic BP < 95 and diastolic BP < 65.
* Adequate intraoperative fluid loading: a minimum of 1500 ml IV fluids should be infused during procedure: at least 300 cc/15 minutes.

Exclusion Criteria:

* Blood coagulopathies resulting in a hypocoagulable state (hemophilia, von Willebrand disease, etc.)
* Blood coagulopathies resulting in a hypercoagulable state (factor V leiden, antithrombin III deficiency, protein C deficiency, protein S deficiency)
* Patients on anti-coagulants (coumadin, plavix, pradaxa, heparin)
* Congestive Heart Failure (at least one medication to treat congestive heart failure)
* Coronary artery disease (s/p bypass, stent or AMI)
* Kidney insufficiency (creatinine > 1.5)
* Aortic or mitral valve disease
* Pulmonary hypertension
* Revision Knee Surgery
* Inadequate intravenous fluid substitution during the procedure 1.5L during 60 minutes.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for primary total knee arthroplasty who meet the qualifications will be consented prior to the surgery.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2014-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Boettner, MD, Principal Investigator — Associate Professor of Orthopaedic Surgery
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anesthesia
Started | 35
Completed | 32
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Anesthesia
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: years] | 66 [44 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Hemoglobin (in g/dl) Levels
Description: To investigate the effect of intraoperative fluid substitution during HEA on hemoglobin levels during and after primary TKA.
Time Frame: up to 48 hours after surgery
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Anesthesia
Number analyzed (Participants) | 32
g/dl
  15 min | 12.2 (1.2)
  30 min | 12.0 (1.2)
  45 min | 11.9 (1.595)
  60 min | 11.8 (1.3)
  PACU stay | 12.0 (1)
  POD1 (24hr) | 11.6 (1.2)
  POD2 (48hr) | 11.0 (1.3)

2. Primary Outcome: Hematocrit (g/dL) Levels
Description: To Investigates the effect of intraoperative fluid substitution during HEA on hematocrit levels during and after primary TKA.
Time Frame: Up to 48 hours after surgery
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Anesthesia
Number analyzed (Participants) | 32
g/dl
  15 min | 36.8 (3.2)
  30 min | 36 (3.1)
  45 min | 35.4 (2.9)
  60 min | 34.7 (3.1)
  PACU | 35.1 (2.7)
  POD1 (24hr) | 35.3 (3.4)
  POD (48hr) | 32.6 (3.2)

ADVERSE EVENTS:
Time Frame: 2 days following surgery
Arm/Group | Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes